CLINICAL TRIAL: NCT00441727
Title: A Randomized, Double-blind, Parallel-group, Multicentre, Phase III Study to Assess the Effect of Esomeprazole 20 or 40 mg od Versus Placebo on the Occurrence of Peptic Ulcers During 26 Weeks in Subjects on Continuous Low Dose Acetylsalicylic Acid (ASA)
Brief Title: Study of Esomeprazole 20 mg or 40 mg vs Placebo Effectiveness on the Occurrence of Peptic Ulcers in Subjects on Low Dose Acetylsalicylic Acid (LDA)
Acronym: Oberon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D961FC00003; EudraCT No. 2006-005073-22
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Gastric Ulcer; Duodenal Ulcer
Keywords: Peptic ulcer; low-dose ASA
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Peptic Ulcer | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Esomeprazole 40 mg (Experimental): Esomeprazole 40 mg
  Interventions: Drug: Esomeprazole 40 mg
- Esomeprazole 20 mg (Experimental): Esomeprazole 20 mg
  Interventions: Drug: Esomeprazole 20 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole 40 mg — Esomeprazole 40 mg once daily
  Arms: Esomeprazole 40 mg
Drug: Esomeprazole 20 mg — Esomeprazole 20 mg once daily
  Arms: Esomeprazole 20 mg
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effect of esomeprazole 20 or 40 mg once daily versus placebo on the occurrence of peptic ulcers during 26 weeks in subjects on continuous low-dose acetylsalicylic acid.

ELIGIBILITY:
Inclusion Criteria:

* Daily intake of low-dose Aspirin (ASA) - The subject must fulfill at least one of the following (a-e):
* Aged ≥65 years.
* Aged ≥18 years and with a documented history of uncomplicated peptic ulcer(s).
* Aged ≥60 years and naïve to low-dose ASA (ie, treatment started within 1 month prior to randomization).
* Aged ≥60 years and with stable coronary artery disease.
* Aged ≥60 years and with complaints of upper gastrointestinal (GI) symptoms that, as judged by the investigator, requires an Esophagogastroduodenoscopy (EGD) and with the finding of ≥5 gastric and/or duodenal erosions at the baseline endoscopy.

Exclusion Criteria:

* Peptic ulcer(s) at baseline esophagogastroduodenoscopy (EGD).
* Reflux esophagitis Los Angeles (LA) classification grade C or D at baseline
* History of peptic ulcer complications such as clinically significant bleeding and/or perforation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2426 (Actual)
Dates: Start 2007-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tore Lind, MD, PhD, Study Director — AstraZeneca; James Scheiman, MD, Principal Investigator — University of Michigan
Locations (189):
- United States (55):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Lancaster, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Carlos, California
  - Research Site, San Diego, California
  - Research Site, Torrington, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Miami, Florida
  - Research Site, New Smyrna Beach, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Plantation, Florida
  - Research Site, South Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Fulton, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Hollywood, Maryland
  - Research Site, Prince Frederick, Maryland
  - Research Site, Brockton, Massachusetts
  - Research Site, Jackson, Mississippi
  - Research Site, Las Vegas, Nevada
  - Research Site, Egg Harbor, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Great Neck, New York
  - Research Site, Fayetteville, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Centerville, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Guthrie, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Cranston, Rhode Island
  - Research Site, Johnston, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Ogden, Utah
  - Research Site, Burke, Virginia
  - Research Site, Chesapeake, Virginia
  - Research Site, Christiansburg, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Milwaukee, Wisconsin
- Argentina (7):
  - Research Site, Capital Federal, Buenos Aires
  - Research Site, Loma Hermosa, Buenos Aires
  - Research Site, Lomas de Zamora, Buenos Aires
  - Research Site, Buenos Aires, Buenos Aires- Argentina
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Mendoza
  - Research Site, Rosario
- Australia (7):
  - Research Site, Caboolture, Queensland
  - Research Site, Carina Heights, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Ballarat, Victoria
  - Research Site, Box Hill, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, NSW
- Bulgaria (5):
  - Research Site, Chirpan
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Canada (17):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Carbonear, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Niagara Falls, Ontario
  - Research Site, North York, Ontario
  - Research Site, Tillsonburg, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Laval
  - Research Site, Longueuil
  - Research Site, Québec
- Czechia (10):
  - Research Site, Beroun
  - Research Site, Brno
  - Research Site, Liberec
  - Research Site, Litoměřice
  - Research Site, Ostrava - Trebovice
  - Research Site, Podbořany
  - Research Site, Poobram
  - Research Site, Prague
  - Research Site, Praha 4 - Sporilov
  - Research Site, Tábor
- Finland (6):
  - Research Site, Jakobstad
  - Research Site, Joensuu
  - Research Site, Mikkeli
  - Research Site, Tampere
  - Research Site, Turku
  - Research Site, Vantaa
- Germany (12):
  - Research Site, Bochum
  - Research Site, Dresden
  - Research Site, Ludwigshafen
  - Research Site, Lüdenscheid
  - Research Site, Magdeburg
  - Research Site, München
  - Research Site, Oelde
  - Research Site, Potsdam
  - Research Site, Rodgau-dudenhofen
  - Research Site, Siegen
  - Research Site, Wangen
  - Research Site, Wolmirstedt
- Indonesia (4):
  - Research Site, Jakarta
  - Research Site, Semarang
  - Research Site, Surabaya
  - Research Site, Yogyakarta
- Mexico (5):
  - Research Site, México, D.f.
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, D.F
  - Research Site, Mexico City
- Norway (13):
  - Research Site, Asker
  - Research Site, Bergen
  - Research Site, Elverum
  - Research Site, Gjøvik
  - Research Site, Hamar
  - Research Site, Levanger
  - Research Site, Lysaker
  - Research Site, Oslo
  - Research Site, Osteros
  - Research Site, Paradis
  - Research Site, Stavanger
  - Research Site, Tromsø
  - Research Site, Ølesund
- Philippines (2):
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (14):
  - Research Site, Bydgoszcz
  - Research Site, Chojnice
  - Research Site, Chrzanów
  - Research Site, Czechowice-Dziedzice
  - Research Site, Częstochowa
  - Research Site, Elblog
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Iława
  - Research Site, Kościerzyna
  - Research Site, Krakow
  - Research Site, Sopot
  - Research Site, Tczew
  - Research Site, Warsaw
- Portugal (8):
  - Research Site, Angra Do Herosmo
  - Research Site, Braga
  - Research Site, Castelo Branco
  - Research Site, Coimbra
  - Research Site, Covilha
  - Research Site, Lisbon
  - Research Site, Setúbal
  - Research Site, Vila Real
- Romania (5):
  - Research Site, Brasov, Brașov County
  - Research Site, Iași, Iaşi
  - Research Site, Bucharest
  - Research Site, Satu Mare
  - Research Site, Tg. Mures
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Slovakia (10):
  - Research Site, Banska Bysterica
  - Research Site, Bánovce nad Bebravou
  - Research Site, Brastislava
  - Research Site, Liptovský Mikuláš
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Nové Mesto nad Váhom
  - Research Site, Piešťany
  - Research Site, Považská Bystrica
  - Research Site, Trnava
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
- South Korea (2):
  - Research Site, Seongnam-si, Kyeonggi-do
  - Research Site, Seoul
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Chiang Mai

REFERENCES:
- [Derived] Scheiman JM, Herlitz J, Veldhuyzen van Zanten SJ, Lanas A, Agewall S, Naucler EC, Svedberg LE, Nagy P. Esomeprazole for prevention and resolution of upper gastrointestinal symptoms in patients treated with low-dose acetylsalicylic acid for cardiovascular protection: the OBERON trial. J Cardiovasc Pharmacol. 2013 Mar;61(3):250-7. doi: 10.1097/FJC.0b013e31827cb626. PMID 23188121
- [Derived] Scheiman JM, Devereaux PJ, Herlitz J, Katelaris PH, Lanas A, Veldhuyzen van Zanten S, Naucler E, Svedberg LE. Prevention of peptic ulcers with esomeprazole in patients at risk of ulcer development treated with low-dose acetylsalicylic acid: a randomised, controlled trial (OBERON). Heart. 2011 May;97(10):797-802. doi: 10.1136/hrt.2010.217547. Epub 2011 Mar 17. PMID 21415072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was randomized 22 February 2007 and last subject completed 28 August 2008. Cardiologists, primary care physicians and gastroenterologists were the primary target investigators.
Groups:
- Esomeprazole 40: Esomeprazole 40 mg every day for 26 weeks in subjects on continuous low-dose ASA (acetylsalicyclic acid) (75-325 mg)
- Esomeproazole 20: Esomeprazole 20 mg every day for 26 weeks in subjects on continuous low dose ASA (75-325 mg)
- Placebo: Placebo every day for 26 weeks in subjects on continuous low-dose ASA (75-325 mg)
Period: Overall Study
Arm/Group | Esomeprazole 40 | Esomeproazole 20 | Placebo
Started | 817 (ITT/randomised) | 804 (ITT/randomised) | 805 (ITT/randomised)
Completed | 711 (ITT/randomised) | 686 (ITT/randomised) | 637 (ITT/randomised)
Not Completed | 106 | 118 | 168
Not completed — Protocol Violation | 19 | 28 | 32
Not completed — Adverse Event | 26 | 33 | 28
Not completed — Lack of Efficacy | 7 | 8 | 48
Not completed — Withdrawal by Subject | 40 | 34 | 47
Not completed — Lost to Follow-up | 5 | 6 | 5
Not completed — Safety Reasons | 3 | 1 | 3
Not completed — Various reason specified | 6 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole 40 | Esomeproazole 20 | Placebo | Total
Number analyzed (Participants) | 817 | 804 | 805 | 2426
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 240 | 246 | 260 | 746
  >=65 years | 577 | 558 | 545 | 1680
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 380 | 375 | 402 | 1157
  Male | 437 | 429 | 403 | 1269

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced the Occurence of Peptic Ulcer(s).
Description: The occurrence of ulcer (mucosal break measuring >= 3 mm over its largest diameter with a sharply demarcated margin) was determined by endoscopy performed at baseline, 8 weeks and 26 weeks or upon withdrawal.
Time Frame: During 26 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole 40 | Esomeproazole 20 | Placebo
Number analyzed (Participants) | 817 | 804 | 805
percentage of participants | 1.35 | 1 | 6.58

2. Secondary Outcome: Percentage of Participants Who Experienced the Occurence of Gastric Ulcer.
Description: The occurrence of gastric ulcer (mucosal break measuring >= 3 mm over its largest diameter with a sharply demarcated margin) was determined by endoscopy performed at baseline, 8 weeks and 26 weeks or upon withdrawal.
Time Frame: During 26 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole 40 | Esomeproazole 20 | Placebo
Number analyzed (Participants) | 817 | 804 | 805
percentage of participants | 1.1 | 0.75 | 4.1

3. Secondary Outcome: Percentage of Participants Who Experienced the Occurrence of Duodenal Ulcer.
Description: The occurrence of duodenal ulcer (mucosal break measuring >= 3 mm over its largest diameter with a sharply demarcated margin) was determined by endoscopy performed at baseline, 8 weeks and 26 weeks or upon withdrawal.
Time Frame: During 26 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole 40 | Esomeproazole 20 | Placebo
Number analyzed (Participants) | 817 | 804 | 805
percentage of participants | 0.24 | 0.25 | 2.73

4. Secondary Outcome: Number of Participants Reporting 0 in the Dichotomized RDQ (Reflux and Disease Questionnaire) Score (0 Versus >0) for the Dyspepsia Dimension During the 26-week Visit or the Week Prior to the Last Visit.
Description: RDQ contains 12 items on a 6-point Likert scale. Six items concern the frequence ('Did not have' to 'Daily') and six items concern the severity ('Did not have' to 'Severe'). The dyspepsia dimension contains the items 'Burning feeling in the center of the upper stomach' and 'Pain in the center of the upper stomach'. Best score possible 0, worst score possible - daily occurrence.
Time Frame: RDQ was assessed at baseline, 8 weeks, 16 week, 26 weeks or upon withdrawal.
Population: Patients randomized who took at least one dose of study drug and completed RDQ questionnaire at baseline and at week 26 or the week prior to last visit were analyzed.
Measure: Number; unit: participants
Groups:
- Esomeprazole 40 mg: Esomeprazole 40 mg every day for 26 weeks in subjects on continuous low-dose ASA (acetylsalicyclic acid) (75-325 mg)
- Esomeprazole 20 mg: Esomeprazole 20 mg every day for 26 weeks in subjects on continuous low-dose ASA (acetylsalicyclic acid) (75-325 mg)
- Placbo: Placebo every day for 26 weeks in subjects on continuous low-dose ASA (acetylsalicyclic acid) (75-325 mg)
Arm/Group | Esomeprazole 40 mg | Esomeprazole 20 mg | Placbo
Number analyzed (Participants) | 782 | 758 | 763
participants | 591 | 577 | 504

5. Secondary Outcome: Number of Participants Reporting 0 in the Dichotomized RDQ (Reflux and Disease Questionnaire) Score (0 Versus >0) for the Gastroesophageal Reflux Disease Dimension During the 26-week Visit or the Week Prior to the Last Visit.
Description: RDQ contains 12 items on a 6-point Likert scale. Six items concern the frequency ('Did not have' to 'Daily') and six items concern the severity ('Did not have' to 'Severe'). Gastroesophageal reflux disease (GERD) items: 'Acid taste in the mouth', 'Unpleasant movement of materials upward from the stomach', 'Burning feeling behind the breastbone' and 'Pain behind the breastbone'. Best score possible 0, worst score possible - daily occurrence.
Time Frame: RDQ was assessed at baseline, 8 weeks, 16 week, 26 weeks or upon withdrawal.
Population: as for outcome 4
Measure: Number; unit: participants
Groups:
- Esomeproazole 20 mg: Esomeprazole 20 mg every day for 26 weeks in subjects on continuous low dose ASA (acetylsalicyclic acid) (75-325 mg)
- Placebo: Placebo every day for 26 weeks in subjects on continuous low-dose ASA (acetylsalicyclic acid) (75-325 mg)
Arm/Group | Esomeprazole 40 mg | Esomeproazole 20 mg | Placebo
Number analyzed (Participants) | 782 | 758 | 763
participants | 554 | 537 | 451

6. Secondary Outcome: Number of Participants With Gastric and/or Duodenal Erosions.
Time Frame: The number of erosions was determined by endoscopy performed at baseline, 8 weeks and 26 weeks or upon withdrawal.
Population: Patients randomized who had endoscopy performed at baseline, 8 weeks and 26 weeks or upon withdrawal.
Measure: Number; unit: participants
Arm/Group | Esomeprazole 40 | Esomeproazole 20 | Placebo
Number analyzed (Participants) | 772 | 753 | 748
participants | 214 | 213 | 380

ADVERSE EVENTS:
Description: Nine (9) randomized subjects were not evaluable for safety analysis because they were never exposed to investigational product. Three (3) additional subjects were excluded from safety. They were exposed to investigational product, but did not have any post-dose data.
Arm/Group | Esomeprazole 40 | Esomeproazole 20 | Placebo
Serious Adverse Events (participants affected / at risk) | 46 | 40 | 35
Other Adverse Events (participants affected / at risk) | 32 | 42 | 31
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Esomeprazole 40 | Esomeproazole 20 | Placebo
Acute Coronary Syndrome (Cardiac disorders) | 0/814 | 1/799 | 0/801
Angina Pectoris (Cardiac disorders) | 2/814 | 0/799 | 1/801
Angina Unstable (Cardiac disorders) | 2/814 | 0/799 | 0/801
Atrial Fibrillation (Cardiac disorders) | 0/814 | 1/799 | 1/801
Cardiac Arrest (Cardiac disorders) | 0/814 | 2/799 | 1/801
Cardiac Failure (Cardiac disorders) | 0/814 | 1/799 | 1/801
Cardiac Failure Congestive (Cardiac disorders) | 1/814 | 0/799 | 0/801
Coronary Artery Disease (Cardiac disorders) | 2/814 | 1/799 | 1/801
Coronary Artery Stenosis (Cardiac disorders) | 0/814 | 0/799 | 1/801
Myocardial Infarction (Cardiac disorders) | 1/814 | 1/799 | 0/801
Myocardial Ischaemia (Cardiac disorders) | 1/814 | 0/799 | 0/801
Vertigo (Ear and labyrinth disorders) | 0/814 | 1/799 | 0/801
Acromegaly (Endocrine disorders) | 0/814 | 0/799 | 1/801
Abdominal Pain (Gastrointestinal disorders) | 1/814 | 0/799 | 0/801
Abdominal Pain Upper (Gastrointestinal disorders) | 1/814 | 0/799 | 0/801
Colitis (Gastrointestinal disorders) | 0/814 | 1/799 | 0/801
Diarrhoea (Gastrointestinal disorders) | 0/814 | 1/799 | 0/801
Diverticulum (Gastrointestinal disorders) | 0/814 | 0/799 | 1/801
Duodenal Perforation (Gastrointestinal disorders) | 0/814 | 1/799 | 0/801
Dyspepsia (Gastrointestinal disorders) | 1/814 | 0/799 | 0/801
Gastric Ulcer (Gastrointestinal disorders) | 0/814 | 0/799 | 1/801
Gastritis (Gastrointestinal disorders) | 1/814 | 0/799 | 0/801
Inguinal Hernia (Gastrointestinal disorders) | 2/814 | 0/799 | 1/801
Intestinal Ischaemia (Gastrointestinal disorders) | 1/814 | 0/799 | 0/801
Intestinal Obstruction (Gastrointestinal disorders) | 0/814 | 1/799 | 0/801
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1/814 | 1/799 | 0/801
Pancreatitis (Gastrointestinal disorders) | 0/814 | 1/799 | 0/801
Pancreatitis Acute (Gastrointestinal disorders) | 2/814 | 1/799 | 0/801
Subileus (Gastrointestinal disorders) | 1/814 | 0/799 | 0/801
Vomiting (Gastrointestinal disorders) | 1/814 | 1/799 | 0/801
Chest Pain (General disorders) | 0/814 | 1/799 | 0/801
Death (General disorders) | 0/814 | 1/799 | 0/801
Non-Cardiac Chest Pain (General disorders) | 1/814 | 0/799 | 1/801
Sudden Death (General disorders) | 1/814 | 0/799 | 0/801
Cholecystitis (Hepatobiliary disorders) | 0/814 | 0/799 | 1/801
Cholecystitis Acute (Hepatobiliary disorders) | 1/814 | 1/799 | 0/801
Cholelithiasis (Hepatobiliary disorders) | 0/814 | 1/799 | 0/801
Hepatitis Toxic (Hepatobiliary disorders) | 0/814 | 1/799 | 0/801
Bronchitis (Infections and infestations) | 0/814 | 1/799 | 0/801
Diverticulitis (Infections and infestations) | 1/814 | 0/799 | 0/801
Erysipelas (Infections and infestations) | 1/814 | 0/799 | 0/801
Lobar Pneumonia (Infections and infestations) | 0/814 | 1/799 | 0/801
Meningitis (Infections and infestations) | 0/814 | 0/799 | 1/801
Pyelonephritis (Infections and infestations) | 1/814 | 0/799 | 0/801
Pyelonephritis Acute (Infections and infestations) | 1/814 | 0/799 | 0/801
Sepsis (Infections and infestations) | 1/814 | 0/799 | 0/801
Urinary Tract Infection (Infections and infestations) | 0/814 | 0/799 | 1/801
Arthropod Bite (Injury, poisoning and procedural complications) | 1/814 | 0/799 | 0/801
Dislocation Of Joint Prosthesis (Injury, poisoning and procedural complications) | 0/814 | 0/799 | 1/801
Femur Fracture (Injury, poisoning and procedural complications) | 0/814 | 0/799 | 1/801
Hand Fracture (Injury, poisoning and procedural complications) | 0/814 | 0/799 | 1/801
Humerus Fracture (Injury, poisoning and procedural complications) | 0/814 | 0/799 | 1/801
Joint Dislocation (Injury, poisoning and procedural complications) | 1/814 | 0/799 | 0/801
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0/814 | 0/799 | 1/801
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1/814 | 0/799 | 0/801
Wrist Fracture (Injury, poisoning and procedural complications) | 0/814 | 0/799 | 1/801
Diabetes Mellitus (Metabolism and nutrition disorders) | 0/814 | 1/799 | 0/801
Gout (Metabolism and nutrition disorders) | 1/814 | 0/799 | 0/801
Hypokalaemia (Metabolism and nutrition disorders) | 0/814 | 1/799 | 0/801
Hyponatraemia (Metabolism and nutrition disorders) | 0/814 | 1/799 | 0/801
Arthritis (Musculoskeletal and connective tissue disorders) | 0/814 | 1/799 | 1/801
Back Pain (Musculoskeletal and connective tissue disorders) | 1/814 | 0/799 | 0/801
Flank Pain (Musculoskeletal and connective tissue disorders) | 0/814 | 0/799 | 1/801
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/814 | 0/799 | 0/801
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0/814 | 0/799 | 1/801
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/814 | 0/799 | 1/801
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/814 | 0/799 | 1/801
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/814 | 0/799 | 1/801
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/814 | 0/799 | 1/801
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/814 | 0/799 | 1/801
Lentigo Maligna Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/814 | 1/799 | 0/801
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/814 | 1/799 | 0/801
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/814 | 1/799 | 1/801
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/814 | 0/799 | 0/801
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/814 | 0/799 | 0/801
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/814 | 0/799 | 1/801
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/814 | 1/799 | 0/801
Signet-Ring Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/814 | 0/799 | 0/801
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/814 | 1/799 | 0/801
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/814 | 0/799 | 1/801
Carotid Arteriosclerosis (Nervous system disorders) | 0/814 | 0/799 | 1/801
Cerebral Circulatory Failure (Nervous system disorders) | 0/814 | 1/799 | 0/801
Cerebral Infarction (Nervous system disorders) | 0/814 | 1/799 | 0/801
Cerebrovascular Accident (Nervous system disorders) | 1/814 | 2/799 | 0/801
Dizziness (Nervous system disorders) | 0/814 | 0/799 | 1/801
Syncope (Nervous system disorders) | 1/814 | 1/799 | 0/801
Transient Ischaemic Attack (Nervous system disorders) | 0/814 | 2/799 | 0/801
Nephrolithiasis (Renal and urinary disorders) | 1/814 | 0/799 | 0/801
Renal Failure Acute (Renal and urinary disorders) | 1/814 | 0/799 | 0/801
Benign Prostatic Hyperplasia (Renal and urinary disorders) | 1/814 | 0/799 | 0/801
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/814 | 0/799 | 0/801
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/814 | 1/799 | 0/801
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/814 | 1/799 | 0/801
Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0/814 | 1/799 | 0/801
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0/814 | 1/799 | 0/801
Deep Vein Thrombosis (Vascular disorders) | 1/814 | 0/799 | 0/801
Hypertensive Crisis (Vascular disorders) | 0/814 | 0/799 | 1/801
Thromboangiitis Obliterans (Vascular disorders) | 0/814 | 0/799 | 1/801
Varicose Vein (Vascular disorders) | 1/814 | 0/799 | 0/801
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Esomeprazole 40 | Esomeproazole 20 | Placebo
Diarrhoea (Gastrointestinal disorders) | 21/814 | 26/799 | 18/801
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 11/814 | 16/799 | 13/801

LIMITATIONS AND CAVEATS:
Not enough patients had peptic ulcer, gastric ulcer, or duodenal ulcer to report the intended primary endpoint of time to peptic ulcer and two secondary endpoints, time to gastric ulcer and time to duodenal ulcer. Percentage used instead.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other